CLINICAL TRIAL: NCT03161691
Title: Perfusion and Collateral Imaging Using C-arm Computed Tomography in the Neuro-Angiography Suite
Brief Title: Perfusion and Collaterals Imaging With C-arm CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Vitor Pereira, Associate Professor of Radiology and Surgery, University Health Network, Toronto
Other Study IDs: TWH -Ver. 3.0 March 17 2017
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic Stroke: Percutaneous neurovascular treatment of acute ischemic stroke patients.
  Interventions: Procedure: Percutaneous treatment of ischemic stroke

INTERVENTIONS:
Procedure: Percutaneous treatment of ischemic stroke — An additional C-arm CT imaging scan will be done during neurovascular treatment to evaluate perfusion and collateral vessels in ischemic stroke patients.

SUMMARY:
Single-center, single-arm pilot study to evaluate the ability of C-arm computed tomography imaging to assess perfusion parameters, collateral vessels, recanalization and brain ischemia in patients with suspected or proven ischemic stroke or brain ischemia in the neuro-angiography suite.

DETAILED DESCRIPTION:
In neurovascular disease, and stroke in particular, physicians often want to be able to detect regions of ischemia in the brain and the recanalization status of cerebral blood vessels. Perfusion and collateral vessel imaging is a possible approach for doing this. These imaging techniques are able to differentiate ischemic core in parenchymal tissue in the brain versus salvageable penumbra tissue around the core. Also the recanalization status of blood vessels can be evaluated using this technique. This study wishes to investigate if the x-ray C-arm in the treatment room can generate perfusion and collateral images of clinical value during treatment, using a technique known as C-arm computed tomography. If this study shows that to be the case, then it might be feasible in the future to bypass CT or MR perfusion/collateral imaging for some patients when they arrive at the hospital, since all this imaging can be done in the treatment room. In the future, this imaging approach may have the potential to simplify and improve patient workflows and reduce the time between hospital arrival and treatment for these patients and could also potentially compensate for missing imaging information.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has suspected or proven ischemic stroke or brain ischemia.
2. Subject requires diagnostic and/or interventional imaging in the neuro-angiography suite.
3. Subject or subject's legally authorized representative has signed an institutionally approved research informed consent form.
4. Subject ≥ 18 years old.

Exclusion Criteria:

1. Subject or subject's legally authorized representative is unable or unwilling to consent to the study.
2. Subject with documented contrast medium injection contraindication due to severe kidney disease or allergy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or proven ischemic stroke or brain ischemia who require diagnostic and/or interventional imaging in the neuro-angiography suite.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinically valuable CACT perfusion images based on a 5-point Likert scale | 1 year
  C-arm computed tomography acquisition perfusion/collateral protocols that provide sufficient image quality to be able to assess ischemic brain perfusion, recanalization and ischemic regions effectively. A 5-point Likert scale questionnaire will be used to evaluate image quality. Cerebral blood volume measurements will also be calculated by image processing software.

SECONDARY OUTCOMES:
Number of participants with CACT perfusion images of comparable quality to standard imaging modalities based on a 5-point Likert scale | 1 year
  CACT perfusion imaging and collateral vessel imaging protocols that are comparable in quality to other standard-of-care imaging modalities (such as CT) that are used for these purposes. A 5-point Likert scale questionnaire will be used to compare the imaging modalities. Cerebral blood volume measurements will also be evaluated based on image processing software calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Pereira, MD, Principal Investigator — University Health Network - Toronto Western Hospital
Locations (1):
- Toronto Western Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No